CLINICAL TRIAL: NCT05582057
Title: Strengths to Grow Preteen: An Online Parenting Resource
Brief Title: Strengths to Grow - Preteen: An Online Parenting Resource
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Margaret Lumley, Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-08-001-2
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Intervention Model Description: The current study is a two-wave randomized controlled trial that employs a 2 (group - between participants) by 2 (time - within participants) mixed measures design to assess a brief online strength-based parenting program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Behavioral: Strengths to Grow Program In an online, self-directed format, the Strengths to Grow: Preteen program will present the principles of strength-based parenting using videos, pictures, reflection questions, and written text. The intervention will communicate that a) every child has a unique set of strengths and that b) noticing and developing these strengths can enhance child and family well-being. It will also provide concrete steps that parents can follow to talk with their child about strengths, and it will provide ideas for family activities that would allow family members to express strengths. Participants will be invited to respond to reflection questions at various points throughout the program.
  Interventions: Behavioral: Strengths to Grow: Preteen
- Waitlist Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Strengths to Grow: Preteen — An online, strength based parenting program for parents of preteens (aged 9-14).
  Arms: Experimental Group

SUMMARY:
Research suggests that strength-based parenting programs can enhance family well-being, but the current formats of these programs (e.g., in-person workshops) are not accessible to many families. The first aim of the study is to adapt Strengths to Grow, an accessible and engaging strength-based parenting program, for pre-teens. The second aim of the study is to assess the effectiveness this adapted program (Strengths to Grow: Preteen). Toward this end, parents of children in Grades 4 through 8 will be invited to complete a brief, online survey of well-being before and a few weeks after completing the online program to assess its impact on well-being.

DETAILED DESCRIPTION:
Strength-based Parenting Strength-based parenting is a style of caregiving which identifies and cultivates strengths in the child and caregiver. When parents employ a strength-based parenting style, youth tend to demonstrate greater academic achievement, resilience, and overall well-being, and parents tend to experience more well-being within the caregiving role. Additionally, it is believed that caregivers can develop a strength-based parenting style through training and practice. For these reasons, several strength-based parenting programs have been developed.

Character Strengths Strength-based parenting programs typically focus on helping parents to identify and develop a particular type of strength known as character strengths. Character strengths are personal qualities that are widely regarded as morally good (e.g., bravery, curiosity, kindness). In 2004, Peterson and Seligman completed a comprehensive review that identified 24 character strengths. The development and use of these 24 character strengths has consistently demonstrated associations with well-being across the lifespan.

Strength-based Parenting Programs The content of strength-based parenting programs typically revolves around introducing parents to character strengths, helping parents to identify character strengths within themselves and their child, teaching parents to notice and encourage their child's use of strengths, and helping parents to employ their strengths within the caregiving role. Within the published literature, strength-based parenting programs have been delivered in two formats: in-person workshops and online handouts. These programs have demonstrated positive effects, including improving caregiving self-efficacy, positive emotions toward the child, and family well-being relative to waitlist control groups. However, the format of these programs may have limited the number of parents who could access and engage with the resources.

Access and Engagement It is important to consider the extent to which caregivers can access and engage with programs because access and engagement are necessary pre-requisites to program effectiveness. Research on parenting programs suggests that in-person workshops are not accessible to many families, particularly families of lower socio-economic status. Online handouts may be more accessible, but may struggle to engage families, as interactive, media-rich online materials tend to be more engaging. To address these concerns, O'Byrne et al (in press) developed an online strength-based parenting intervention for kindergarten-aged children, Strengths to Grow, designed to maximize accessibility and engagement by providing the program online using interactive rather than static materials.

An Online, Interactive, Strength-based Parenting Program for Preteens In a preliminary evaluation of the Strengths to Grow program, O'Byrne et al. (in press) found that parents reacted positively to the online, interactive format and the strength-based content. Additionally, within the sample, the program was accessible to families of lower socio-economic status who are difficult to access with in-person resources. While a more formal assessment of the effectiveness of Strengths to Grow is underway, preliminary findings suggest that the Strengths to Grow model may be effective at engaging hard-to-reach parents. However, the current Strengths to Grow program is designed specifically for parents of kindergarten to Grade 3 children. Because the strengths profiles and displays of kindergarten children may be different from other age groups, the current iteration of Strengths to Grow may not be generalizable to older children. Thus, the present research seeks to broaden the reach of Strengths to Grow by adapting it for parents of pre-adolescents (Grades 4 to 8; Strengths to Grow: Preteen). In addition, the present study will investigate 1. who is accessing Strengths to Grow: Preteen; 2. how Strengths to Grow: Preteen is being accessed; 3. whether participants report being satisfied with Strengths to Grow: Preteen; and 4. whether specific participant characteristics predict satisfaction with Strengths to Grow: Preteen.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child(ren) who is enrolled in Grade 4 to 8 at the Upper Grand District School Board in Guelph, Ontario
* Able to read and write in English (linguistic proficiency equivalent to a Grade 8 reading level or greater)
* Consent to participate in the research study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Parenting Sense of Competence Scale: Efficacy Subscale (Johnston & Mash, 1989) | 1 week
  Caregiving Self-Efficacy; 1 = Strongly Disagree to 6 = Strongly Agree; higher scores indicate increased sense of competence
Modified Differential Emotions Scale (Fredrickson, 2013) [Instructions modified to capture child-oriented emotions consistent with Waters and Sun (2016)] | 1 week
  Parent child-Oriented Positive Emotions; 0 = Never to 4 = Most of the time; higher scores indicate increased positive emotions
Subjective Happiness Scale (Lyubomirsky & Lepper, 1999) | 1 week
  Parent happiness; 1 to 7 (various anchors); higher scores indicated increased happiness
Patient Health Questionnaire 4 (Kroenke et al., 2009) [Instructions modified to capture parent's perceptions of child mental health] | 1 week
  Child mental health; 0 = Not at all to 4 = Nearly every day; higher scores indicate worse mental health
Perceived Stress Scale (Cohen, 1994) | 1 week
  Parent stress; 0 = Never to 4 = Very often; higher scores indicate higher stress

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lumley, PhD, CPsych, Principal Investigator — University of Guelph
Locations (1):
- Upper Grand District School Board, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data as this has not been approved by our Research Ethics Board.

REFERENCES:
- [Background] Friedmann, J. (2022). Assessing Character Strengths in Young Children (Doctoral dissertation, University of Guelph).
- [Background] Danaher BG, Boles SM, Akers L, Gordon JS, Severson HH. Defining participant exposure measures in Web-based health behavior change programs. J Med Internet Res. 2006 Aug 30;8(3):e15. doi: 10.2196/jmir.8.3.e15. PMID 16954125
- [Background] Eisner M, Meidert U. Stages of parental engagement in a universal parent training program. J Prim Prev. 2011 Apr;32(2):83-93. doi: 10.1007/s10935-011-0238-8. PMID 21424399
- [Background] Fernandez MA, Eyberg SM. Predicting treatment and follow-up attrition in parent-child interaction therapy. J Abnorm Child Psychol. 2009 Apr;37(3):431-41. doi: 10.1007/s10802-008-9281-1. PMID 19096926
- [Background] Fredrickson, B. L. (2013). Chapter One-Positive Emotions Broaden and Build. In P. Devine & A. Plant (Eds.), Advances in Experimental Social Psychology (Vol. 47, pp. 1-53). Academic Press. https://doi.org/10.1016/B978-0-12-407236-7.00001-2
- [Background] Ivtzan, I., Niemiec, R. M., & Briscoe, C. (2016). A study investigating the effects of Mindfulness-Based Strengths Practice (MBSP) on wellbeing. International Journal of Wellbeing, 6(2), 1- 13. https://doi.org/10/gfscgj
- [Background] Jach, H. K., Sun, J., Loton, D., Chin, T.-C., & Waters, L. (2018). Strengths and subjective wellbeing in adolescence: Strengthbased parenting and the moderating effect of mindset. Journal of Happiness Studies, 19(2), 567-586. https://doi.org/10/gfscg9
- [Background] Johnston, C., & Mash, E. J. (1989). A Measure of Parenting Satisfaction and Efficacy. Journal of Clinical Child Psychology, 18(2), 167-175. https://doi.org/10.1207/s15374424jccp1802_8
- [Background] Kazdin, A. E., & Rabbitt, S. M. (2013). Novel models for delivering mental health services and reducing the burdens of mental illness. Clinical Psychological Science, 1(2), 170-191. https://doi.org/10/gc4pnm
- [Background] Lavigne JV, Lebailly SA, Gouze KR, Binns HJ, Keller J, Pate L. Predictors and correlates of completing behavioral parent training for the treatment of oppositional defiant disorder in pediatric primary care. Behav Ther. 2010 Jun;41(2):198-211. doi: 10.1016/j.beth.2009.02.006. Epub 2009 Dec 5. PMID 20412885
- [Background] Lyubomirsky, S., & Lepper, H. S. (1999). A Measure of Subjective Happiness: Preliminary Reliability and Construct Validation. Social Indicators Research, 46(2), 137-155. https://doi.org/10.1023/A:1006824100041
- [Background] McGoron, L., & Ondersma, S. J. (2015). Reviewing the need for technological and other expansions of evidence-based parent training for young children. Children and Youth Services Review, 59, 71-83. https://doi.org/10/f8bhbv
- [Background] O'Byrne R, Thompson R, Friedmann JS, Lumley MN. Parent Engagement with an Online, School-Based, Character Strengths Promotion Program. Int J Appl Posit Psychol. 2022;7(3):355-377. doi: 10.1007/s41042-022-00072-4. Epub 2022 Aug 11. PMID 35971433
- [Background] Peterson, C., & Seligman, M. E. P. (2004). Introduction to a manual of the sanities. In Character strengths and virtues (pp.18-104). American Psychological Association; Oxford University Press. https://books.scholarsportal.info/uri/ebooks/ebooks0/oxford/2009- 11-30/3/0195167015
- [Background] Ritterband, L. M., Cox, D. J., Gordon, T. L., Borowitz, S. M., Kovatchev, B. P., Walker, L. S., & Sutphen, J. L. (2006). Examining the Added Value of Audio, Graphics, and Interactivity in an Internet Intervention for Pediatric Encopresis. Children's Health Care, 35(1), 47-59. https://doi.org/10.1207/s15326888chc3501_5
- [Background] Shoshani A, Shwartz L. From Character Strengths to Children's Well-Being: Development and Validation of the Character Strengths Inventory for Elementary School Children. Front Psychol. 2018 Nov 2;9:2123. doi: 10.3389/fpsyg.2018.02123. eCollection 2018. PMID 30450070
- [Background] Waters, L. (2015a). The relationship between strength-based parenting with children's stress levels and strength-based coping approaches. Psychology, 06(06), 689-699. https://doi.org/10/gdj4w6
- [Background] Waters, L. (2015b). Strength-based parenting and life satisfaction in teenagers. Advances in Social Sciences Research Journal, 2(11), 158-173. https://doi.org/10.14738/assrj.211.1651
- [Background] Waters, L. (2020). Using positive psychology interventions to strengthen family happiness: A family systems approach. The Journal of Positive Psychology, 0(0), 1-8. https://doi.org/10.1080/17439760.2020.1789704
- [Background] Waters, L., Loton, D., & Jach, H. K. (2018). Does Strength-Based Parenting Predict Academic Achievement? The Mediating Effects of Perseverance and Engagement. Journal of Happiness Studies. https://doi.org/10/gfscg8
- [Background] Waters, L., & Sun, J. (2016). Can a brief strength-based parenting intervention boost self-efficacy and positive emotions in parents? International Journal of Applied Positive Psychology, 1(1), 41-56. https://doi.org/10/gfschb